CLINICAL TRIAL: NCT02033213
Title: Intraoperative Volume Restriction in Esophageal Carcinoma Surgery: an Exploratory Randomized Clinical Trial
Brief Title: Volume Restriction in Esophageal Carcinoma Surgery: Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klinički Bolnički Centar Zagreb (Other)
Responsible Party: Principal Investigator, Maja Karaman Ilić, MD PhD, Klinički Bolnički Centar Zagreb
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: JORTK3
Record Dates: First submitted 2014-01-07; First posted 2014-01-10 (Estimated); Results first posted 2014-05-26 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-04

CONDITIONS: Esophageal Neoplasm
Keywords: intraoperative; fluid management; esophageal carcinoma; surgery; gas exchange; tissue perfusion
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Restrictive group (Active Comparator): Patients who received ≤ 8ml/kg/h of intraoperative fluid. A fluid administered during surgery: Plasma-Lyte 148 (pH 7.4; Viaflo, Baxter, US), 10% Aminoven (Fresenius Kabi AG, Bad Homburg, Germany) at 0.5 ml/kg/h, 5 ml/kg of colloid (6% Voluven 130/0.4, Fresenius Kabi AG, Bad Homburg, Germany), packed red blood cells.
  Interventions: Other: Restrictive group
- Liberal group (Active Comparator): Patients who received > 8 ml/kg/h of fluid. A fluid used during surgery: Plasma-Lyte 148 (pH 7.4; Viaflo, Baxter, US), 10% Aminoven (Fresenius Kabi AG, Bad Homburg, Germany) at 0.5 ml/kg/h, 5 ml/kg of colloid (6% Voluven 130/0.4, Fresenius Kabi AG, Bad Homburg, Germany), packed red blood cells.
  Interventions: Other: Liberal group

INTERVENTIONS:
Other: Restrictive group — A group of patients who received ≤ 8ml/kg/h of intraoperative fluid during esophageal carcinoma surgery.
  The fluid administered: Plasma-Lyte 148 (pH 7.4; Viaflo, Baxter, US), 10% Aminoven (Fresenius Kabi AG, Bad Homburg, Germany) at 0.5 ml/kg/h, 5 ml/kg of colloid (6% Voluven 130/0.4, Fresenius Kabi AG, Bad Homburg, Germany), packed red blood cells.
  Other Names: Intraoperative restrictive fluid management
  Arms: Restrictive group
Other: Liberal group — A group of patients who received > 8 ml/kg/h of intraoperative fluid during esophageal carcinoma surgery.
  The fluid admnistered: Plasma-Lyte 148 (pH 7.4; Viaflo, Baxter, US), 10% Aminoven (Fresenius Kabi AG, Bad Homburg, Germany) at 0.5 ml/kg/h, 5 ml/kg of colloid (6% Voluven 130/0.4, Fresenius Kabi AG, Bad Homburg, Germany), packed red blood cells.
  Other Names: Intraoperative liberal fluid management
  Arms: Liberal group

SUMMARY:
An exploratory single-centre randomized clinical trial was performed in order to investigate whether the fluid volume administered during esophageal carcinoma surgery affects pulmonary gas exchange and tissue perfusion.

DETAILED DESCRIPTION:
A convenience sample of 16 patients admitted to the Department of Thoracic surgery University Hospital Centre Zagreb and scheduled for esophageal carcinoma surgery were enrolled prospectively in the study between June 2011 and August 2012.

Patients were randomly allocated into two groups, one of which received ≤ 8ml/kg/h of intraoperative fluid ("restrictive group") and another that received > 8 ml/kg/h of fluid ("liberal group").

Patients were excluded if they were younger than 18 years; if they had severe lung disease, chronic renal insufficiency, or a physical status classification > III on the American Society of Anesthesiologists (ASA) scale; or if it was impossible to perform epidural catheter placement or thoraco-phreno-laparotomy.

All patients underwent esophagectomy carried out according to the Lewis-Tanner approach.

Data on arterial oxygen partial pressure (PaO2), inspired oxygen fraction (FiO2), and the ratio PaO2/FiO2 were collected 10 min after anesthesia was induced and again 6 h after surgery. Data on the metabolic markers creatinine and lactate were collected 10 min after anesthesia induction and 6 h after surgery.

ANOVA tests were performed to determine significant differences in mean values between study groups. Independent-sample t-tests were used to test differences in mean values between the restrictive and liberal groups for each of the two sets of measurements separately (10 minutes after anesthesia induction and 6 hr after surgery). P < 0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* esophageal carcinoma
* Lewis Tanner procedure (median laparotomy and right thoracotomy)

Exclusion Criteria:

* younger than 18 years
* severe lung disease
* chronic renal insufficiency
* a physical status classification > III on the American Society of Anesthesiologists (ASA) scale
* impossible to perform epidural catheter placement
* thoraco-phreno-laparotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maja Karaman Ilić, MD PhD, Principal Investigator — Clinical Hospital Centre Zagreb
Locations (1):
- Department of Thoracic surgery "Jordanovac" University Hospital Centre Zagreb, Zagreb, City of Zagreb, Croatia

REFERENCES:
- [Derived] Karaman Ilic M, Madzarac G, Kogler J, Stancic-Rokotov D, Hodoba N. Intraoperative volume restriction in esophageal cancer surgery: an exploratory randomized clinical trial. Croat Med J. 2015 Jun;56(3):290-6. doi: 10.3325/cmj.2015.56.290. PMID 26088854

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Restrictive Group | Liberal Group
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Restrictive Group | Liberal Group | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.91 (8.31) | 52.41 (13.41) | 53.12 (1.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 6 | 4 | 10
ASA score [Mean (Standard Deviation); unit: units on a scale] — The American Society of Anesthesiologists (ASA) Physical Status classification system consists of six categories, as described below:
  ASA PS 1: Normal healthy patient. ASA PS 2: Patients with mild systemic disease. ASA PS 3: Patients with severe systemic disease. ASA PS 4: Patients with severe systemic disease that is a constant threat to life. ASA PS 5: Moribund patients who are not expected to survive without the operation. ASA PS 6: A declared brain-dead patient who organs are being removed for donor purposes.
  Smaller number is better.
  units on a scale | 2.61 (0.51) | 2.75 (0.46) | 2.71 (0.48)
Body weight [Mean (Standard Deviation); unit: kg] | 70.01 (18.91) | 66.31 (12.61) | 68.11 (17.61)

OUTCOME MEASURES:

1. Primary Outcome: Pulmonary Gas Exchange During and After Esophageal Carcinoma Surgery (PaO2/FiO2 Ratio)
Description: At the given time point, 10 minutes after beginning of the Lewis Tanner procedure and 6 hours after, arterial oxygen partial pressure (PaO2), inspired oxygen fraction (FiO2), and the PaO2/FiO2 ratio will be measured. The results of Pa02/FiO2 ratio will be compared between two groups for each time point separately.
Time Frame: 10 minutes, 6 hours
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Restrictive Group | Liberal Group
Number analyzed (Participants) | 8 | 8
mmHg
  10 minutes | 345.01 (35.31) | 330.11 (34.71)
  6 hours | 315.51 (32.91) | 307.11 (30.31)
Statistical Analysis 1: Comparison: Restrictive Group vs Liberal Group; The measurement was assessed at 10 minutes time point; Test type: Superiority or Other; p = 0.410, t-test, 1 sided — P < 0.05 was considered significant
Statistical Analysis 2: Comparison: Restrictive Group vs Liberal Group; The measurement was assessed at 6 hours time point; Test type: Superiority or Other; p = 0.621, t-test, 1 sided — P < 0.05 was considered significant

2. Primary Outcome: Creatinine Values During and After Esophageal Carcinoma Surgery
Description: At the given time points, 10 minutes after beginning of the Lewis Tanner procedure and 6 hours after, creatinine blood levels will be measured. The results will be compared between two groups for each time point separately.
Time Frame: 10 minutes, 6 hours
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Restrictive Group | Liberal Group
Number analyzed (Participants) | 8 | 8
μmol/L
  10 minutes | 91.91 (12.67) | 90.88 (14.99)
  6 hours | 93.51 (16.37) | 100.88 (18.33)
Statistical Analysis 1: Comparison: Restrictive Group vs Liberal Group; The measurement was assessed at 10 minutes time point; Test type: Superiority or Other; p = 0.791, t-test, 1 sided — P < 0.05 was considered significant
Statistical Analysis 2: Comparison: Restrictive Group vs Liberal Group; The measurement was assessed at 6 hours time point; Test type: Superiority or Other; p = 0.410, t-test, 1 sided — P < 0.05 was considered significant

3. Primary Outcome: Lactate Values During and After Esophageal Carcinoma Surgery
Description: At the given time points, ten minutes after beginning of the Lewis Tanner procedure and six hours after procedure, blood levels of the lactate will be measured and compared between two groups for each time point separately.
Time Frame: 10 minutes, 6 hours
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Restrictive Group | Liberal Group
Number analyzed (Participants) | 8 | 8
mmol/L
  10 minutes | 3.93 (1.33) | 3.26 (1.25)
  6 hours | 2.69 (0.91) | 2.40 (1.08)
Statistical Analysis 1: Comparison: Restrictive Group vs Liberal Group; The measurement aws assessed at 10 minutes time point; Test type: Superiority or Other; p = 0.322, t-test, 1 sided — P < 0.05 was considered significant
Statistical Analysis 2: Comparison: Restrictive Group vs Liberal Group; The measurement was assessed at 6 hours time point; Test type: Superiority or Other; p = 0.574, t-test, 1 sided — P < 0.05 was considered significant

4. Primary Outcome: Changes in Lactate Levels During Esophageal Carcinoma Surgery Using Restrictive or Liberal Fluid Management.
Description: At the given time points, ten minutes after beginning of the Lewis Tanner procedure and six hours after procedure, blood levels of the lactate will be measured and compared inside the same group (liberal or restrictive).
Time Frame: 10 minutes, 6 hours
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Restrictive Group | Liberal Group
Number analyzed (Participants) | 8 | 8
mmol/L
  10 minutes | 3.93 (1.33) | 3.26 (1.25)
  6 hours | 2.69 (0.91) | 2.40 (1.08)
Statistical Analysis 1: Comparison: Restrictive Group; Test type: Superiority or Other; p = 0.030, t-test, 1 sided — P < 0.05 was considered significant
Statistical Analysis 2: Comparison: Liberal Group; Test type: Superiority or Other; p = 0.096, t-test, 1 sided — P < 0.05 was considered significant

5. Secondary Outcome: Duration of Surgery
Description: Total time of Lewis-Tanner procedure will be measured and compared between two groups.
Time Frame: End of surgery.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Restrictive Group: Patients who received ≤ 8ml/kg/h of intraoperative fluid. A fluid administered during surgery: Plasma-Lyte 148 (pH 7.4; Viaflo, Baxter, US), 10% Aminoven (Fresenius Kabi AG, Bad Homburg, Germany) at 0.5 ml/kg/h, 5 ml/kg of colloid (6% Voluven 130/0.4, Fresenius Kabi AG, Bad Homburg, Germany), packed red blood cells.
  Restrictive group: A group of patients who received ≤ 8ml/kg/h of intraoperative fluid during esophageal carcinoma surgery.
  The fluid administered: Plasma-Lyte 148 (pH 7.4; Viaflo, Baxter, US), 10% Aminoven (Fresenius Kabi AG, Bad Homburg, Germany) at 0.5 ml/kg/h, 5 ml/kg of colloid (6% Voluven 130/0.4, Fresenius Kabi AG, Bad Homburg, Germany), packed red blood cells.
- Liberal Group: Patients who received > 8 ml/kg/h of fluid. A fluid used during surgery: Plasma-Lyte 148 (pH 7.4; Viaflo, Baxter, US), 10% Aminoven (Fresenius Kabi AG, Bad Homburg, Germany) at 0.5 ml/kg/h, 5 ml/kg of colloid (6% Voluven 130/0.4, Fresenius Kabi AG, Bad Homburg, Germany), packed red blood cells.
  Liberal group: A group of patients who received > 8 ml/kg/h of intraoperative fluid during esophageal carcinoma surgery.
  The fluid admnistered: Plasma-Lyte 148 (pH 7.4; Viaflo, Baxter, US), 10% Aminoven (Fresenius Kabi AG, Bad Homburg, Germany) at 0.5 ml/kg/h, 5 ml/kg of colloid (6% Voluven 130/0.4, Fresenius Kabi AG, Bad Homburg, Germany), packed red blood cells.
Arm/Group | Restrictive Group | Liberal Group
Number analyzed (Participants) | 8 | 8
minutes | 275.61 (91.21) | 324.41 (116.61)
Statistical Analysis 1: Comparison: Restrictive Group vs Liberal Group; Test type: Superiority or Other; p = 0.362, t-test, 1 sided

6. Secondary Outcome: Total Volume of Administered Intraoperative Fluid
Description: Total volume of intraoperatively given fluid according to the protocol will be measured and compared between two groups.
Time Frame: End of surgery
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Restrictive Group | Liberal Group
Number analyzed (Participants) | 8 | 8
milliliters | 2823.75 (965.8) | 3960.00 (755.9)
Statistical Analysis 1: Comparison: Restrictive Group vs Liberal Group; Test type: Superiority or Other; p = 0.020, t-test, 1 sided

ADVERSE EVENTS:
Arm/Group | Restrictive Group | Liberal Group
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

LIMITATIONS AND CAVEATS:
Small number of participants due to small overall number of patients with esophageal cancer treated in our hospital.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No